CLINICAL TRIAL: NCT05717374
Title: Efficacy and Safety of Methylprednisolone Versus Dexamethasone in Caudal Block for Children Undergoing Hypospadias Surgical Repair: A Bi-center Randomized Controlled Study
Brief Title: Methylprednisolone Versus Dexamethasone in Pediatric Caudal Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammed Alseoudy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.22.12.1971.R1
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Caudal Block

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: The study subjects and the resident assessing the outcomes will be blinded to the study group. A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Dexamethasone (Active Comparator): will receive 0.5 ml/kg volume (bupivacaine 0.25 % + dexamethasone 0.1mg/kg) for caudal block
  Interventions: Drug: caudal block using dexamethasone
- Group Methylprednisolone (Experimental): will receive 0.5 ml/kg volume (bupivacaine 0.25% + methylprednisolone 0.5mg/kg) for caudal block
  Interventions: Drug: caudal block using methylprednisolone

INTERVENTIONS:
Drug: caudal block using dexamethasone — patient will receive 0.5 ml/kg volume (bupivacaine 0.25 % + dexamethasone 0.1mg/kg) through the sacral hiatus
  Other Names: caudal dexamethasone
  Arms: Group Dexamethasone
Drug: caudal block using methylprednisolone — patients will receive 0.5 ml/kg volume (bupivacaine 0.25% + methylprednisolone 0.5mg/kg) through the sacral hiatus
  Other Names: caudal methylprednisolone
  Arms: Group Methylprednisolone

SUMMARY:
This randomized, double-blind, controlled bi-center study was designed to compare the postoperative analgesic efficacy of dexamethasone and methylprednisolone in caudal block for children undergoing hypospadias surgical repair using the duration of analgesia as the primary outcome. We hypothesize that methylprednisolone will provide superior postoperative analgesia than dexamethasone when added to bupivacaine for caudal block. This study will be conducted on 80 male patients of American Society of Anesthesiologists physical status I-II of with their age ranging from 1 to 6 years scheduled for surgical repair of hypospadias. The patients will be randomly assigned into 2 groups:- Group D: will receive 0.5 ml/kg volume (bupivacaine 0.25 % + dexamethasone 0.1mg/kg) Group M: will receive 0.5 ml/kg volume (bupivacaine 0.25% + methylprednisolone 0.5mg/kg) The main collected data will be the duration of analgesia (first need for rescue analgesia ), the severity of postoperative pain according to FLACC and the side effects like nausea and vomiting, respiratory depression.

DETAILED DESCRIPTION:
Hypospadias repair surgery is an invasive surgery that results in significant postoperative pain. pain alters the quality of life and satisfaction of the patients and results in manipulation of wounds, infection, bleeding, and wound dehiscence leading to unfavorable surgical outcome .

As a plan for postoperative pain prophylaxis in children, different analgesic techniques have been used as preemptive analgesia such as local infiltration of anesthesia, penile block, epidural block and caudal block in addition to general anesthesia. Caudal block is found to be one of most succeeded technique in hypospadias repair and decreases the postoperative analgesia consumption.

Bupivacaine is a local anesthetic commonly used via caudal epidural route but gives limited duration of analgesia. Therefore, the addition of other drugs in an attempt to improve the quality and duration of analgesia given by bupivacaine has been studied.

Examples of additives drugs used in the caudal epidural are opioids, alpha 2 agonist as dexmedtomidine and clonidine which produce prolongation of the duration of the analgesia, but their undesirable effect may limit its use as nausea, vomiting, pruritus, urinary retention and respiratory depression.

Epidural corticosteroids have a long history of safe and effective use in the treatment of low back and radicular pain due to their strong anti-inflammatory effect encouraging use in management of acute postoperative pain.

In pediatric surgical patients presenting for mainly lower abdominal surgery, a meta-analysis revealed clinically meaningful prolongation of the duration of analgesia from caudal blockade by adjuvant dexamethasone versus placebo. In addition to doubling to tripling the duration of analgesia, adjuvant dexamethasone has a rescue analgesia sparing effect and reduces post postoperative nausea and vomiting.

A vast majority of literature supports the efficacy of particulate steroids like methylprednisolone over dexamethasone in providing longer analgesia in management of chronic pain conditions.

Aim of the work and hypothesis:

To the best of our knowledge, this is the first study that will evaluate the analgesic efficacy and safety of caudal methylprednisolone in pediatric patients. This randomized, double-blind, controlled bi-center study was designed to compare the postoperative analgesic efficacy of dexamethasone and methylprednisolone in caudal block for children undergoing hypospadias surgical repair using the duration of analgesia as the primary outcome. The investigators hypothesize that methylprednisolone will provide superior postoperative analgesia than dexamethasone when added to bupivacaine for caudal block.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* American Society of Anesthesiologists physical status I-II of
* age ranging from 1 to 6 years
* scheduled for surgical repair of hypospadias

Exclusion Criteria:

* a history of neurodevelopmental delay
* type I diabetes
* coagulopathy
* known allergy to any local anesthetic or steroid,
* known congenital anomaly of the spine and local infection.

Ages: 1 Year to 6 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
duration of analgesia | Up to 24 hours after the procedure]
  first need for rescue analgesia will be recorded

SECONDARY OUTCOMES:
the severity of postoperative pain according to FLACC score | Up to 24 hours after the procedure]
  Pain levels will be assessed post operatively using the 10-point behavioral face, leg, activity, cry, consolability (FLACC) pain scale, with a minimum score of 0 and a maximum of 10 at 0,1, 2, 4, 6, 12, 24 hours
side effects | Up to 24 hours after the procedure]
  side effects including nausea and vomiting, respiratory depression, hyperglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No